CLINICAL TRIAL: NCT03203135
Title: Assesment of the Impact of a Nutritional Prevention Programme for Employees in Staggered Hours.
Acronym: PREV'HODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Professor, Institut Pasteur de Lille
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A00812-51
Record Dates: First submitted 2017-06-19; First posted 2017-06-29 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Shift-work; Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Nutritional prevention programme
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Nutritional prevention programme — The nutritional prevention programme will offer a wide range of food and physical activity activities adapted to the life of the company (example: culinary demonstration, physical activity, provision of fruit baskets, etc.) .
  Arms: Intervention Group

SUMMARY:
Staggered work affects about 20% of French employees and its health risks are now well known. They concern physical health (sleep disorders, weight gain, cancer, cardiovascular disorders, nutritional problems, etc.) and psychological health. Faced with these "alarming" findings, it is necessary to find ways of improvement and levers of action to prevent them.

This project aims to set up and evaluate a nutritional health prevention programme for the benefit of employees in staggered hours from CITEO. CITEO is a company of social mediation.

The objectives of the project are twofold: to evaluate the impact of working conditions in shifted schedules on food behavior and on to improve their eating behaviors.

How? Focusing on the pleasure of eating through a nutritional prevention program in which various and varied actions will be proposed but always adapted to the life of the company (example: culinary demonstration, physical activity, provision of baskets of Fruits, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Participants working at CITEO in staggered hours

Exclusion Criteria:

* Pregnant woman, person with severe pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 14 months
  in centimeters
Weight | 14 months
  in kg
Blood pressure | 14 months
  in mm Hg
Metabolic parameters (Total cholesterol, HDL, LDL, Triglycerdies, glycemia) | 14 months
  in g/l
Food consumption behavior and food representations | 14 months
  score
Physical activity level | 14 months
  Ricci and gagnon score
Height | 14 months
  in meters

SECONDARY OUTCOMES:
Motivation to change habits | 14 months
  scale of Prochaska
Body Feeling | 14 months
  Analog visual scales (AVS)
Well-being | 14 months
  AVS
Stress | 14 months
  AVS
Sleep quality | 14 months
  AVS
Fatigue | 14 months
  scale of Pichot

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — IPL
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France